CLINICAL TRIAL: NCT03772145
Title: TOUR: Tofacitinib Response in Ulcerative Colitis - a Real World Prospective Multi-center Study
Brief Title: Tofacitinib Response in Ulcerative Colitis - a Real World Prospective Multi-center Study
Acronym: TOUR
Status: Terminated | Type: Observational
Why Stopped: Futility; recruitment to slow to justify longer study duration
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-2435
Record Dates: First submitted 2018-12-04; First posted 2018-12-11 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Inflammatory bowel diseases; Tofacitinib
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Tofacitinib: Adult patients, age 18 years or older, with UC, who within 2 weeks have been started on tofacitinib therapy for moderate to severe UC or who plan to start this therapy within the next 2 weeks. The start of the tofacitinib therapy must have been or be initiated in the setting of standard of care therapy

SUMMARY:
The overarching goal of this study, is to create a longitudinally followed, well phenotyped cohort of patients with UC starting treatment with tofacitinib in the setting of standard of care who have linked clinical data and self-reported outcome data that will lead to evaluation of efficacy and safety of tofacitinib in the real-life setting. The specific aims for the study are:

1. Create a prospective cohort of well phenotyped (proctitis vs. rectosigmoiditis vs. extensive) adult UC patients with serial clinical and patient-reported data collected throughout the course of 12 months of tofacitinib therapy. Enrolled patients on therapy will be followed up to 36 months after the start of therapy.
2. To determine clinical response rates and persistence of therapy with tofacitinib for induction and maintenance therapy
3. Describe the incidence of specific drug-associated adverse events (shingles, serious infections), hospitalizations and surgeries in the standard of care setting.
4. Assess the correlation of various outcome measures in ulcerative colitis (Simple Clinical Colitis Activity Index (SCCAI), partial Mayo index, 6-point index) and endoscopic outcomes via the endoscopic Mayo Score

DETAILED DESCRIPTION:
The proposed prospective tofacitinib registry is a prospective patient cohort with the goal of evaluating the efficacy and safety of this drug in "real life". All patients starting tofacitinib for ulcerative colitis in the setting of standard of care therapy will be eligible within of 4 weeks of start of therapy. Preferentially, patients will be enrolled at the visit where therapy is initiated. At baseline patient characteristics including extent of disease, previous therapies (including number of previously failed biologics) and pro-inflammatory laboratory markers (CRP, if available calprotectin) will be captured in a prospective web-based database. Additionally, each consented study participant will be enrolled in a web-based prospective patient powered registry (PPR) to evaluate patient report outcomes (PRO's) (such as validated measures for depression, social satisfaction, pain, fatigue) and safety events (e.g. hospitalizations; herpes zoster, complications requiring discontinuation of tofacitinib).

The following outcomes will be assessed: Response and remission as assessed by the Simple Clinical Colitis Activity Index (SCCAI) (primary endpoint), in addition secondary outcomes will include: the partial Mayo score, the 6-point subscore of the Mayo score, and the Manitoba index, need for steroids, need for surgery or hospitalization, need for dosing intensification or reduction of dosing as well as persistence of tofacitinib therapy. Endoscopy information will be collected if done as part of routine care, but the study will not have an endoscopic requirement. Sites will be encouraged to report a Mayo endoscopic score if done as part of routine care as a secondary endpoint. The outcomes will be determined in the setting of the standard of care visits, which normally are scheduled at the end of induction (approx. 6-12 weeks after the start of tofacitinib) and during maintenance therapy after 4-6 and 9-12 months and then every 3-4 months up to 36 months. PRO's and safety will be assessed with the PPR instrument at baseline, daily in the first 2 weeks to better understand rapidity of onset, and after 6,10,14,22,30,38,46 and 54 weeks and then every 3-4 months up to 36 months. The analyses of these data will facilitate UC patient care and improve the overall quality of IBD therapy in the US and worldwide. This study is to be conducted according to US and international standards of Good Clinical Practice (FDA Title 21 part 312 and International Conference on Harmonization guidelines), applicable government regulations and Institutional research policies and procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, age 18 years or older, with UC, who within 2 weeks have been started on tofacitinib therapy for moderate to severe UC or who plan to start this therapy within the next 2 weeks. The start of the tofacitinib therapy must have been or be initiated in the setting of standard of care therapy
2. Anticipation that the patient will be followed by the participating center at least for the next 12 months
3. Diagnosis of UC must be established on the basis of standard clinical, radiographic, endoscopic, and histologic criteria as described below.

Exclusion Criteria:

* 1. Patients will be excluded if they meet any of the following criteria:

  1. Inability to provide informed consent
  2. Patients presenting for a one-time consultation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, age 18 years or older, with UC, who within 2 weeks have been started on tofacitinib therapy for moderate to severe UC or who plan to start this therapy within the next 2 weeks. The start of the tofacitinib therapy must have been or be initiated in the setting of standard of care therapy
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2023-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Change in clinical response from baseline | At baseline and at approximately 2, 4, 8, 20 and 52 weeks after start of tofacitinib
  Clinical response as assessed by the Simple Clinical Colitis Activity Index (SCCAI)

SECONDARY OUTCOMES:
Change in clinical remission from baseline | At baseline and at approximately 2, 4, 8, 20 and 52
  Clinical remission as assessed by the Simple Clinical Colitis Activity Index (SCCAI)
Persistence of the initial tofacitinib dose | 12 months
  Persistence of initial tofacitinib dose

CONTACTS AND LOCATIONS:
Overall Officials: Hans Herfarth, MD, Principal Investigator — University of North Carolina; Millie Long, Principal Investigator — University of North Carolina
Locations (1):
- Division of Gastroenterology and Hepatology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is currently no plan to share the anonymized data with other investigators. But this may change in the future

REFERENCES:
- [Result] Long MD, Afzali A, Fischer M, Hudesman D, Abdalla M, McCabe R, Cohen BL, Ungaro RC, Harlan W, Hanson J, Konijeti G, Polyak S, Ritter T, Salzberg B, Seminerio J, English E, Zhang X, Sharma PP, Herfarth HH. Tofacitinib Response in Ulcerative Colitis (TOUR): Early Response After Initiation of Tofacitinib Therapy in a Real-world Setting. Inflamm Bowel Dis. 2023 Apr 3;29(4):570-578. doi: 10.1093/ibd/izac121. PMID 35700276
- [Result] Herfarth HH, Afzali A, Fischer M, Hudesman D, Abdalla M, McCabe R, Cohen BL, Ungaro RC, Harlan W, Hanson J, Konijeti GG, Polyak S, Ritter T, Salzberg B, Seminerio J, English E, Zhang X, Long MD. Clinical Long-Term Outcomes of Patient-Reported Outcomes in the Prospective Real-World Tofacitinib Response in Ulcerative Colitis Registry. Clin Transl Gastroenterol. 2024 Mar 1;15(3):e00669. doi: 10.14309/ctg.0000000000000669. PMID 38131617